CLINICAL TRIAL: NCT01144624
Title: A Phase II, Multicentre, Randomised, Double-Blind, Placebo-Controlled, Dose Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of Intravenous Infusions of AZD9773 (CytoFab™) in Japanese Patients With Severe Sepsis and/or Septic Shock
Brief Title: A Study to Assess Safety,and Tolerability of 2 Doses of AZD9773 (CytoFab™) in Japanese With Severe Sepsis/Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0620C00005
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-09

CONDITIONS: Severe Sepsis; Septic Shock
Keywords: TNF neutralisation
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — AZD9773; CytoFab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AZD9773 250 units/kg (1 infusion) + 50 units/kg (9 infusions) (Dose Cohort 1):
  AZD9773 500 units/kg (1 infusion) + 100 units/kg (9 infusions) (Dose Cohort 2)
  Interventions: Drug: AZD9773
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9773 — A single loading dose followed by 9 maintenance doses; doses to be given every 12 hours over a period of 5 days
  Other Names: CytoFab™
  Arms: 1
Drug: Placebo — Intravenous infusion of a saline solution
  Arms: 2

SUMMARY:
The two co-primary objectives of this study are to assess in Japanese patients with severe sepsis and/or septic shock: 1) the safety and tolerability of two different doses of intravenous AZD9773 and 2) the PK of AZD9773.

The secondary objective is to make a preliminary assessment of the pharmacodynamics of two different doses of intravenous AZD9773 in Japanese patients with severe sepsis and/or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Japanese adults with a first episode of sepsis during this hospitalisation and objective evidence of infection that requires parenteral antibiotics.
* At least 2 of 4 SIRS criteria in the 24 hours before organ dysfunction (must include either fever OR elevated white blood cells [WBC])
* Cardiovascular or respiratory dysfunction.

Exclusion Criteria:

* Immunocompromising comorbidities or concomitant medications:

  1. Advanced human immunodeficiency virus (HIV) infection (CD4 ≤50/mm3).
  2. Haemopoietic or lymphoreticular malignancies not in remission.
  3. Receiving radiation therapy or chemotherapy.
  4. Any organ or bone marrow transplant within the past 24 weeks.
  5. Absolute neutrophil count <500 per μL.
  6. High dose steroids or other immunocompromising drugs.
* Concomitant diseases:

  1. Deep-seated fungal infection or active tuberculosis.
  2. Severe chronic liver disease associated with portal hypertension, cirrhosis, chronic ascites or Child-Pugh class C.
  3. History of chronic hypercarbia, respiratory failure in past 6 months or use of home oxygen in the setting of severe chronic respiratory disease.
  4. Neuromuscular disorders that impact breathing/spontaneous ventilation.
  5. Quadriplegia.
  6. Cardiac arrest in the past 30 days.
  7. New York Heart Association functional Class III or IV due to heart failure or any disorder.
  8. Burns over > 30% of body surface area in the past 5 days.
* Medication and allergy disqualifications.

  1. Treatment with anti-TNF agents within the last 8 weeks.
  2. Previously received ovine derived products (CroFab™, DigiFab™).
  3. Sheep product allergy or allergy to papain, chymopapain.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lindemann, MD, Study Director — AstraZeneca; Wayne Dankner, MD, Study Director — PAREXEL International Medical Services; Warren Botnick, MD, Study Director — PAREXEL International Medical Services
Locations (7):
- Japan (7):
  - Research Site, Sapporo, Hokkaido
  - Research Site, Kobe, Hyōgo
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Osaka, Osaka
  - Research Site, Sumiyoshi-ku, Osaka
  - Research Site, Hachiōji, Tokyo
  - Research Site, Ohta-ku, Tokyo

REFERENCES:
- [Derived] Aikawa N, Takahashi T, Fujimi S, Yokoyama T, Yoshihara K, Ikeda T, Sadamitsu D, Momozawa M, Maruyama T. A Phase II study of polyclonal anti-TNF-alpha (AZD9773) in Japanese patients with severe sepsis and/or septic shock. J Infect Chemother. 2013 Oct;19(5):931-40. doi: 10.1007/s10156-013-0612-y. Epub 2013 May 17. PMID 23681364
- See also: D0620C00005 Study Report Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=241&filename=D0620C00005.pdf
- See also: redacted-CSP-D0620C00005.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=241&filename=Japan_Ph2b_D0620C00005_redacted_text_18_July-2014.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at six centres in Japan.
Groups:
- Dose Cohort 1: AZD9773 250/50 units/kg IV
- Dose Cohort 2: AZD9773 500/100 units/kg IV
- Placebo: Saline
Period: Overall Study
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Placebo
Started | 7 | 7 | 6
Received Treatment | 7 | 7 | 6
Completed Treatment | 7 (One patient died after completing the full course of study treatment.) | 7 | 6 (Two patients died during the dosing period. Death was not a reason for treatment discontinuation.)
Completed | 7 (One patient died during the study. Death was not a reason for treatment or study discontinuation.) | 7 | 6 (Two patients died during the study. Death was not a reason for treatment or study discontinuation.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Placebo | Total
Number analyzed (Participants) | 7 | 7 | 6 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (10.89) | 77.6 (10.45) | 77.7 (17.64) | 75.4 (12.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 11
  Male | 4 | 3 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of AZD9773
Description: Number of patients with treatment-emergent adverse events and number of patients who died over 28 days
Time Frame: 28 day study period
Population: Safety analysis set
Measure: Number; unit: Participants
Groups:
- Arm 1 - Dose Cohort 1: AZD9773 250/50 units/kg IV
- Arm 2 - Dose Cohort 2: AZD9773 500/100 units/kg IV
- Arm 3 - Placebo: Saline
Arm/Group | Arm 1 - Dose Cohort 1 | Arm 2 - Dose Cohort 2 | Arm 3 - Placebo
Number analyzed (Participants) | 7 | 7 | 6
Participants
  Number of Patients with Treatment-Emergent AEs | 7 | 7 | 6
  Number of Patients who Died over 28 days | 1 | 0 | 2

2. Primary Outcome: Pharmacokinetics of AZD9773
Description: Maximum concentration at steady state (Cmax ss) for serum total and specific fabs
Time Frame: From first dose to last dose (Day 5/6 or at premature treatment discontinuation)
Population: Pharmacokinetic analysis set
Measure: Geometric Mean (Full Range); unit: ug/mL
Arm/Group | Arm 1 - Dose Cohort 1 | Arm 2 - Dose Cohort 2 | Arm 3 - Placebo
Number analyzed (Participants) | 7 | 5 | 0
ug/mL
  Cmax ss for serum total fabs | 38.48 [30.5 to 62.4] | 71.04 [41.7 to 90.7] |
  Cmax ss for serum specific fabs | 1.823 [1.31 to 2.62] | 3.335 [1.92 to 4.62] |

3. Secondary Outcome: Pharmacodynamic Effects of AZD9773 on TNF-alpha
Description: TNF-alpha levels over approximately 6 days following the first dose
Time Frame: Levels taken at baseline, over the dosing period (up to Day 5/6)
Population: Safety analysis set
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Arm 1 - Dose Cohort 1 | Arm 2 - Dose Cohort 2 | Arm 3 - Placebo
Number analyzed (Participants) | 7 | 7 | 6
pg/ml
  TNF-alpha level at baseline | 1.000 [0.92 to 8.89] | 1.690 [0.92 to 2.65] | 8.810 [1.13 to 29.17]
  TNF-alpha level 1-2 hours post-first dose | 0.920 [0.92 to 5.93] | 0.990 [0.92 to 2.18] | 7.425 [0.92 to 28.40]
  TNF-alpha level on Day 6 (pre-morning dose) | 1.710 [0.92 to 14.90] | 1.140 [0.92 to 1.57] | 1.560 [0.92 to 3.00]

ADVERSE EVENTS:
Arm/Group | Dose Cohort 1 | Dose Cohort 2 | Placebo
Serious Adverse Events (participants affected / at risk) | 4/7 | 1/7 | 1/6
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort 1 (N=7) | Dose Cohort 2 (N=7) | Placebo (N=6)
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Cohort 1 (N=7) | Dose Cohort 2 (N=7) | Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 1 | 0
Cardiovascular Insufficiency (Cardiac disorders) | 0 | 1 | 0
Mitral Valve Incompetence (Cardiac disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1
Ventricular Extrasystoles (Cardiac disorders) | 1 | 2 | 1
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0
Pyloric Stenosis (Congenital, familial and genetic disorders) | 0 | 1 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0
Conjunctival Hyperaemia (Eye disorders) | 0 | 1 | 0
Conjunctival Oedema (Eye disorders) | 0 | 1 | 0
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 1 | 0 | 0
Anal Erosion (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 3
Gastric Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis Erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Hypomotility (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus Paralytic (Gastrointestinal disorders) | 1 | 2 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Catheter Site Haematoma (General disorders) | 0 | 0 | 1
Device Leakage (General disorders) | 1 | 0 | 0
Disuse Syndrome (General disorders) | 2 | 1 | 1
Fat Necrosis (General disorders) | 1 | 0 | 0
Generalised Oedema (General disorders) | 2 | 0 | 0
Injection Site Erythema (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 2 | 0
Oedema Peripheral (General disorders) | 1 | 3 | 0
Pain (General disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Abdominal Abscess (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis Staphylococcal (Infections and infestations) | 1 | 0 | 0
Colostomy Infection (Infections and infestations) | 1 | 0 | 0
Fungaemia (Infections and infestations) | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 1 | 0
Incision Site Cellulitis (Infections and infestations) | 1 | 0 | 0
Infectious Peritonitis (Infections and infestations) | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 1 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia Bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 2 | 0 | 2
Pseudomembranous Colitis (Infections and infestations) | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1 | 0
Tinea Cruris (Infections and infestations) | 0 | 0 | 1
Tracheostomy Infection (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal Anastomotic Leak (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tracheal Obstruction (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 1 | 0
Blood Pressure Decreased (Investigations) | 1 | 0 | 0
Body Temperature Increased (Investigations) | 0 | 1 | 0
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Heart Rate Increased (Investigations) | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 1 | 0
Pancreatic Enzymes Increased (Investigations) | 0 | 1 | 0
Urine Output Decreased (Investigations) | 0 | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic Alkalosis (Metabolism and nutrition disorders) | 2 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mental Disorder Due To A General Medical Condition (Psychiatric disorders) | 2 | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tracheal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin Erosion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin Haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Vascular Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermabrasion (Surgical and medical procedures) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less